CLINICAL TRIAL: NCT04475185
Title: Interventional, Open, Non-comparative, Multicenter Study to Assess the Safety and Effectiveness of the Use of the MakAir Artificial Ventilator in the Expected Situation of a Shortage of Technical Devices for Invasive Mechanical Ventilation, Linked to the Coronavirus COVID-19
Brief Title: Safety and Effectiveness Assessment of the MakAir Artificial Ventilator
Acronym: COVRESP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Manufacturer's decision following failure of sequence 2. Protocol unadapted to the security and performance evaluation of the new MakAir device capabilities in non-invasive ventilation (NIV).
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: RC20_0173
Record Dates: First submitted 2020-07-15; First posted 2020-07-17 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MakAir (Experimental)
  Interventions: Device: MakAir

INTERVENTIONS:
Device: MakAir — MakAir artificial ventilator

SUMMARY:
The objective of our study is to carry out an evaluation of the safety and the effectiveness of the use of the MakAir respirator as useful supplement in situation of shortage of technical devices of assistance to the mechanical invasive ventilation, related to COVID-19 through a protocol in 3 successive sequences.

ELIGIBILITY:
Inclusion Criteria:

Sequence 1 :

* Patient for whom a certificate has been signed by a support person / family member / close relative independent of the sponsor.
* Adult
* Non-hypoxemic patient (PaO2 / FiO2> 300)
* Patient requiring invasive mechanical ventilation> 24 hours
* Stabilized patient, i.e. not needing an increase in oxygenation for at least 6 hours

Sequence 2 :

* Patient for whom a certificate of consent has been signed by a support person / family member / close relative independent of the sponsor.
* Adult
* Patient with mild to moderate Acute respiratory distress syndrome (300> Pa02 / FiO2> 100)
* Patient requiring invasive mechanical ventilation> 3 days
* Stabilized patient, i.e. having not required an increase in oxygenation for at least 6 hours

Sequence3 :

* Patient for whom a certificate of consent has been signed by a support person / family member / close relative independent of the sponsor or waiver due to life-threatening emergency.
* Adult
* Patient with mild to moderate Acute respiratory distress syndrome (PaO2 / FiO2> 100) or without Acute respiratory distress syndrome
* Patient requiring invasive mechanical ventilation for any duration
* Situation of shortage among centers investigating technical devices for invasive ventilation to treat all patients

Exclusion Criteria:

Sequence 1 and sequence 2:

* Patient positive or showing signs of Covid-19 infection
* Tracheotomized patient
* History of pulmonary emphysema or severe to moderate chronic obstructive pulmonary disease
* Patient in recovery and withdrawal phase of ventilatory assistance
* Pneumothorax or pneumomediastinum
* Hemodynamic instability
* Intracranial hypertension
* Pregnant woman (A urine or blood pregnancy test must be performed for women of childbearing age)
* Major protected (guardianship, curatorship and under the protection of justice)
* Lack of affiliation to the French social security system
* Participation in another interventional clinical trial

Sequence3 :

* Tracheotomized patient
* History of pulmonary emphysema or severe to moderate moderate chronic obstructive pulmonary disease
* Patient in recovery and withdrawal phase of ventilatory assistance
* Pneumothorax or pneumomediastinum
* Hemodynamic instability
* Intracranial hypertension
* Pregnant woman (A urine or blood pregnancy test must be performed for women of childbearing age)
* Major protected (guardianship, curatorship and under the protection of justice)
* Lack of affiliation to the French social security system
* Participation in another interventional clinical trial on mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-12-19 (Actual); Study Completion 2020-12-19 (Actual)

PRIMARY OUTCOMES:
Number of dysfunctions | 24 hours for sequence 1
  Number of dysfunctions which can lead to or have led to "respiratory" adverse events or to serious adverse events (SAE)
Number of dysfunctions | 5 days for sequence 2
  Number of dysfunctions which can lead to or have led to "respiratory" adverse events or to serious adverse events (SAE)
Number of dysfunctions | 10 days for sequence 3
  Number of dysfunctions which can lead to or have led to "respiratory" adverse events or to serious adverse events (SAE)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Roquilly, MD, Study Director — Nantes University Hospital
Locations (2):
- France (2):
  - CHRU Brest, Brest, Finistère
  - CHU Nantes, Nantes, Loire-Atlantique